CLINICAL TRIAL: NCT04386447
Title: Phase II, Multicenter, Open-label, Rct With an Adaptive Design, to Assess Efficacy of Intravenous Administration of Oxytocin in Hospitalized Patients Affected by COVID-19
Brief Title: Phase II RCT to Assess Efficacy of Intravenous Administration of Oxytocin in Patients Affected by COVID-19
Acronym: OsCOVID19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was not approved by the Italian Medicines Agency (AIFA).
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: University of Parma (Other)
Responsible Party: Principal Investigator, Tiziana Meschi, Director of the Geriatric Rehabilitation Medical Department, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OsCOVID19
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Covid-19; Corona Virus Infection; SARS-CoV 2
Keywords: Covid-19; Oxytocin; Corona Virus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Oxytocin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin 40 UI + SOC (Experimental): In addition to standard treatment, patients in the experimental arm will receive intravenous OT with dilution of 40 UI OT in 500cc physiological solution NaCl 9%. OT will be administered with continuous pump infusion with 62,5 ml/h. The clinician will have the option to decrease infusion speed based on significant variations in arterial pressure, otherwise, the total 25 UI or 40 UI amount will be infused in 8 hours. Treatment duration will be 10 days
  Interventions: Drug: Oxytocin
- Oxytocin 25 UI + SOC (Experimental): In addition to standard treatment, patients in the experimental arm will receive intravenous OT with dilution of 25 UI OT in 500cc physiological solution NaCl 9%. OT will be administered with continuous pump infusion with 62,5 ml/h. The clinician will have the option to decrease infusion speed based on significant variations in arterial pressure, otherwise, the total 25 UI or 40 UI amount will be infused in 8 hours. Treatment duration will be 10 days
  Interventions: Drug: Oxytocin
- Standard of Care (Other): Standard of Care (SoC). Standard of Care will comply with the indications of the Emilia-Romagna Region for the treatment of covid-19, and will include the following:
  * Oxygen supply or non-invasive ventilation to target peripheral blood saturation > 94%
  * Hydroxychloroquine 200mg b.i.d w/o an initial 1-2 days loading dose of 400 mg bid for 1-2 days (the dose may be reduced in patients with advanced CKD according to local protocols) or remdesivir 200 mg in.v on day 1, followed by a 100 mg q.d.
  * Antiretroviral therapy (usually for 5 days) with lopinavir / ritonavir or darunavir / cobicistat is permitted
  * Azithromycin 500 mg q.d., usually for 5 days, is permitted in patients with suspected bacterial superinfection, paying particular attention to safety, considering reports of risk of adverse events in association with hydroxychloroquine
  * Prophylaxis for deep vein thrombosis
  * Steroids are not routinely recommended but may be considered in selected patients.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Oxytocin — In addition to standard treatment, patients in the experimental arm will receive intravenous OT with dilution of 25 UI or 40 UI OT in 500cc physiological solution NaCl 9%. OT will be administered with continuous pump infusion with 62,5 ml/h. The clinician will have the option to decrease infusion speed based on significant variations in arterial pressure, otherwise, the total 25 UI or 40 UI amount will be infused in 8 hours. Treatment duration will be 10 days
  Other Names: Oxytocin OT
  Arms: Oxytocin 25 UI + SOC; Oxytocin 40 UI + SOC
Drug: Standard of Care — Standard of Care (SoC). Standard of Care will comply with the indications of the Emilia-Romagna Region for the treatment of covid-19, and will include the following:
  * Oxygen supply or non-invasive ventilation to target peripheral blood saturation > 94%
  * Hydroxychloroquine 200mg b.i.d w/o an initial 1-2 days loading dose of 400 mg bid for 1-2 days (the dose may be reduced in patients with advanced CKD according to local protocols) or remdesivir 200 mg in.v on day 1, followed by a 100 mg q.d.
  * Antiretroviral therapy (usually for 5 days) with lopinavir / ritonavir or darunavir / cobicistat is permitted
  * Azithromycin 500 mg q.d., usually for 5 days, is permitted in patients with suspected bacterial superinfection, paying particular attention to safety, considering reports of risk of adverse events in association with hydroxychloroquine
  * Prophylaxis for deep vein thrombosis
  * Steroids are not routinely recommended but may be considered in selected patients.
  Other Names: SOC
  Arms: Standard of Care

SUMMARY:
Introduction There are currently no treatments with demonstrated efficacy for COVID-19 infection. Epidemiological evidence points to the existence of intrinsic protection factors which make young persons and women more resistant to the infection, whereas older patients with multiple illnesses, above all with heart disease, are at greatest risk. This trial proposes treatment initiated in the early stages of the disease, when clinical worsening is most likely, with intravenous Oxytocin (OT), an endogenous hormone currently safely used in clinical practice. The selection of this molecule is based on numerous experimental and clinical observations, which show its activity in modulating resistance to pathogens, in mitigating overall cardiovascular risk, and in acting on the production of Nitric Oxide (ON) in the lungs, which is emerging as a key therapeutic factor for the improvement of respiratory function in patients with SARS-COVID 19. Finally, OT is physiologically produced by the human body, especially in the female sex and in the age ranges that coincide with most resistant patients. In routine clinical practice, OT exhibits an excellent therapeutic index, in absence of significant adverse effects.

Primary aim To assess the effects of Oxytocin in addition to standard therapy, with respect to Standard of Care (SoC), in reducing the number of patients who enter a critical stage Secondary aim

To describe:

* Mortality 28 days after randomization
* Time to mechanical ventilation during the study
* Duration of dependency on oxygen supply
* Length of stay
* Temporal trend of clinical improvement (7-category ordinal scale)
* Safety analysis

DETAILED DESCRIPTION:
Intervention In addition to standard treatment, patients in the experimental arm will receive intravenous OT with dilution of 25 UI or 40 UI OT in 500cc physiological solution NaCl 9%. OT will be administered with continuous pump infusion with 62,5 ml/h. The clinician will have the option to decrease infusion speed based on significant variations in arterial pressure, otherwise, the total 25 UI or 40 UI amount will be infused in 8 hours. Treatment duration will be 10 days

Standard of Care (SoC). Standard of Care will comply with the indications of the Emilia-Romagna Region for the treatment of covid-19, and will include the following:

* Oxygen supply or non-invasive ventilation to target peripheral blood saturation > 94%
* Hydroxychloroquine 200mg b.i.d w/o an initial 1-2 days loading dose of 400 mg bid for 1-2 days (the dose may be reduced in patients with advanced CKD according to local protocols) or remdesivir 200 mg in.v on day 1, followed by a 100 mg q.d.
* Antiretroviral therapy (usually for 5 days) with lopinavir / ritonavir or darunavir / cobicistat is permitted
* Azithromycin 500 mg q.d., usually for 5 days, is permitted in patients with suspected bacterial superinfection, paying particular attention to safety, considering reports of risk of adverse events in association with hydroxychloroquine
* Prophylaxis for deep vein thrombosis
* Steroids are not routinely recommended but may be considered in selected patients.

Study design Phase II, multicenter, open-label, experimental randomized controlled trial with an adaptive design, aiming to assess superiority of Oxytocin administration vs SoC.

The adaptive design includes Stage 1, which aims to define the more active of the two considered OT doses, verify endpoints, the target population and the necessary sample size for the following Stage. Selection between the two considered doses (25 UI e 40 UI) will be based on the proportion of patients for which one of the conditions that make up the endpoint is recorded (see below). To this end, for each of the 2 dosages of the experimental agent, a single arm, single stage Fleming design will be applied. Patients enrolled in this Stage will be assigned by balanced randomization (1:1) to one of the two OT doses. The decisional algorithm requires that in a sample of 25 patients, at least 20 (80%) do not worsen to a critical stage (main endpoint) with respect to an expected 17 (68%) with only SOC.

In Stage 2, patients in the experimental arm will receive the dose selected in Stage 1. The study, on two parallel groups, will use unbalanced randomization, because patients who received the selected dose in Stage 1 will be included in the experimental arm to achieve equal sample size between the two arms (60+60) for the analysis of final endpoints Sample size Stage 1 - sample is determined according to the single arm single stage Fleming design applied to each of the 2 investigated OT doses (25 and 40 UI). 25 patients for each dose are estimated necessary to demonstrate a statistically significant difference considering the one-tail test with an alpha probability of 10% and a statistical power of 80%.

Stage 2 - determined using as comparison the test for proportions. From available data, it is assumed that during 14 days of hospitalization the proportion of patients in the SoC group who enters a critical stage (primary endpoint) is 30%, versus 12% in the experimental arm. Using a two-tail test, an alpha probability of 10% and a statistical power of 80%, was estimated that 60 patients per arm are necessary to demonstrate a statistically significant difference

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of pneumonia caused by COVID-19
* Respiratory and/or systemic symptoms and initial mild respiratory failure and with objective signs of lung involvement
* Respiratory frequency ≥25/min, blood oxygen saturation (SaO2) < 95% in A-A, PaO2/FiO2 ratio < 300
* Hospital admission since less than 48 hours
* Signature of informed consent for study participation

Exclusion Criteria:

* MEWS score > 4
* Severe multiple organ failure
* Recent cardiomyopathy, unstable angina, acute myocardial infarction
* Severe kidney failure with glomerular filtration rate less than 30 ml/min or renal replacement therapy or peritoneal dialysis
* History of diabetes insipidus or severe hyponatremia (<128 mEq/L) or hypernatremia (>155 mEq/L)
* QT interval which in the opinion of the patient's treating physician contraindicates therapy with OT
* State of shock
* Women who are pregnant or nursing
* Known intolerance or hypersensitivity to the drug or its excipients
* Treatment with antirejection agents
* Individuals with severe liver failure
* Patients enrolled in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of cases who during 14 exhibit one of the following conditions | 14 days
  Proportion of cases who during 14 days exhibit one of the following conditions (the most severe):
  * respiratory failure that requires mechanical ventilation
  * organ failure that requires intensive care monitoring and treatment
  * death

SECONDARY OUTCOMES:
Mortality 28 days after randomization | 28 days
  Mortality 28 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Meschi, MD,PhD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (3):
- CNRS, Lyon, France
- Italy (2):
  - Azienda Ospedaliero Universitaria di Parma, Parma, PR
  - Ospedale San Francesco, Nuoro